CLINICAL TRIAL: NCT00687843
Title: Phase III Randomized Controlled Study of Postoperative Adjuvant Therapy Using TS-1 or TS-1+PSK for Stage II or III Gastric Cancer Patients
Brief Title: Study of TS-1 or TS-1 + PSK for Gastric Cancer Patients
Acronym: TMOG-GC01
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tokyo Metropolitan Oncology Group (Other)
Responsible Party: Principal Investigator, Yoshiaki Iwasaki, M.D., Ph.D., Department of Surgery, Tokyo Metropolitan Cancer and Infectious Disease Center Komagome Hospital., Tokyo Metropolitan Oncology Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMOG-GC01
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; TS-1; PSK; Relapse-free survival
MeSH Terms: conditions — Stomach Neoplasms | interventions — titanium silicide; polysaccharide-K

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): The TS-1 group
  Interventions: Drug: Tegafur-gimeracil-oteracil potassium (TS-1)
- 2 (Experimental): The TS-1+PSK Group
  Interventions: Drug: Tegafur-gimeracil-oteracil potassium (TS-1); Drug: Krestin (PSK)

INTERVENTIONS:
Drug: Tegafur-gimeracil-oteracil potassium (TS-1) — 80 mg/m2, PO from day 1 to day 28 of each 42 day cycle. Number of Cycles: 8
  Other Names: TS-1
Drug: Krestin (PSK) — 3 g, PO from day 1 to day 336
  Other Names: PSK
  Arms: 2

SUMMARY:
Since it is not uncertain about efficacy of combination therapy with PSK and TS-1 in gastric cancer, in this study, we compare efficacy and safety of postoperative adjuvant therapy using TS-1 or TS-1+PSK in the stage II or III gastric cancer patients.

DETAILED DESCRIPTION:
TS-1 is an oral anticancer drug approved in Japan consisting of tegafur (a pro-drug of fluorouracil, 5-FU), gimeracil and oteracil potassium. The response rate of TS-1 in the untreated advanced gastric cancer patients was 44.6% in the late phase II study. In 2007, efficacy of the adjuvant therapy using TS-1 in the resected gastric cancer patients was demonstrated by ACTS-GC study group conducted in Japan. PSK is an oral anticancer drug approved in Japan consisting of protein-bound polysaccharide extracted from mycelium of Trametes (Coriolus) versicolor, a kind of mushroom. Even though survival benefit by PSK in combination with adjuvant chemotherapy using 5-FU or tegafur in the postoperative gastric cancer patients was already demonstrated, it is not uncertain about efficacy of combination therapy with PSK and TS-1 in gastric cancer. In this study, we compare efficacy and safety of postoperative adjuvant therapy using TS-1 or TS-1+PSK in the stage II or III gastric cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient who is pathologically confirmed as gastric cancer
* Patient who has received surgery with D2 or more lymph node dissection and whose final curability of surgical resection is grade A or B
* Patient whose final stage is II (except for T1), IIIA, or IIIB
* Patient without liver, peritoneal and distant metastasis, and who is negative in peritoneal cytological diagnosis
* Patient whose age at the registration is ranging between 20 and 80 years old
* Patient who has not received any preoperative therapy including radiotherapy, chemotherapy and immunotherapy
* Patient who has received surgery for gastric cancer within six weeks before the registration, and is judged to be capable of oral administration
* Patient who has no serious concurrent complications, and satisfies the following criteria

  * White blood cell count: > LLN or > 4,000 /mm3
  * Platelet count: > 100,000 /mm3
  * Serum total bilirubin: < 1.5 mg/dL
  * Serum AST (GOT), ALT (GPT): < 2.5 * ULN
  * Serum creatinine: < ULN
* Patient who has received an explanation of this study by assent documents, and has given written informed consent to participate in this study

Exclusion Criteria:

* Patient with metachronous or synchronous multicancer
* Patient who contraindicates to TS-1
* Patient who requires continuous use of flucytosine, phenytoin or warfarin potassium
* Patient who has experienced serious drug allergy over grade 3 in the past
* Patient with serious complications including paralysis of intestine, ileus, interstitial pneumonitis, fibroid lung, uncontrollable diabetes mellitus, heart insufficiency, renal insufficiency or hepatic insufficiency
* Patient with diarrhea (watery stool)
* Patient who is pregnant or in lactation, or wish to become pregnant during this study
* Male patient who intends to make someone pregnant during this study
* Patient with HIV positive
* Patient who is judged to be inappropriate as subject to this study by the principal investigator or the doctors in charge

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2008-06; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival | Five years after surgery

SECONDARY OUTCOMES:
Overall survival, quality of life, drug compliance, adverse events, serial changes of tumor markers | Five years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Masatsugu Kitamura, MD, Study Chair
Locations (1):
- Tokyo Metropolitan Cancer and Infectious Disease Center Komagome Hospital, Tokyo, Tokyo, Japan

REFERENCES:
- [Background] Sakuramoto S, Sasako M, Yamaguchi T, Kinoshita T, Fujii M, Nashimoto A, Furukawa H, Nakajima T, Ohashi Y, Imamura H, Higashino M, Yamamura Y, Kurita A, Arai K; ACTS-GC Group. Adjuvant chemotherapy for gastric cancer with S-1, an oral fluoropyrimidine. N Engl J Med. 2007 Nov 1;357(18):1810-20. doi: 10.1056/NEJMoa072252. PMID 17978289
- [Background] Nakazato H, Koike A, Saji S, Ogawa N, Sakamoto J. Efficacy of immunochemotherapy as adjuvant treatment after curative resection of gastric cancer. Study Group of Immunochemotherapy with PSK for Gastric Cancer. Lancet. 1994 May 7;343(8906):1122-6. doi: 10.1016/s0140-6736(94)90233-x. PMID 7910230